CLINICAL TRIAL: NCT06970652
Title: Virtual Reality Intervention for Stress Reduction Among Young Adults
Brief Title: Virtual Reality (VR) for Stress Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City University of New York, School of Public Health (Other)
Collaborators: MindCo Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0338-PHHP
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-04

CONDITIONS: Stress; Resilience; Quality of Life; Depressive Symptoms; Anxiety; Sleep; Physical Activity
Keywords: virtual reality; young adults; stress; stress management
MeSH Terms: conditions — Depression; Anxiety Disorders; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention)
- Intervention (Experimental): MindCo Relief, a mobile VR-based stress management application
  Interventions: Device: virtual reality

INTERVENTIONS:
Device: virtual reality — Participants in the intervention group received access to the MR smartphone application and a smartphone-compatible VR headset, both developed by MindCo Health.32 The application contained a stress reduction program that comprised a structured sequence of 77 modules designed to be completed over the course of 8 weeks. Each module was designed to be completed in approximately 7 minutes, and each module needed to be completed before progressing to the next module. Forty modules used VR, and for these modules, participants placed their personal smartphones running the MR application in the VR headset, and the smartphone provided all audiovisual content. All other modules used smartphones without the VR headset.
  Arms: Intervention

SUMMARY:
This is a randomized pilot trial that aims to examine the impact of smartphone-based Virtual Reality (VR) intervention, MindCo Relief, in reducing stress levels and perceived anxiety, depression, and quality of life among young adults.

DETAILED DESCRIPTION:
Research has shown that young adults are more likely to experience high stress levels due to the combined pressures of academic achievement, career development, financial strain, and navigating interpersonal relationships. High stress levels may contribute to sleep disturbances, anxiety, and depressive symptoms. While cognitive-behavioral therapy (CBT) and mindfulness-based stress reduction (MBSR) have shown effectiveness, traditional interventions are not always accessible or appealing to young adults due to barriers such as stigma, availability, or personal preference.

This study aims to assess the feasibility and preliminary efficacy of MindCo Relief, a mobile virtual reality (VR)-based stress management program. The study will recruit 70 young adults aged 18-29 residing in New York City who report moderate to high perceived stress based on the Perceived Stress Scale (PSS-10). Participants must own a smartphone (iOS or Android), be able to operate the study app, and not be enrolled in other stress reduction programs or have photosensitive epilepsy. After online eligibility screening and signed the informed consent, participants will visit the City University of New York Graduate School of Public Health and Health Policy (CUNY SPH) for baseline assessments, hair sample collection, and equipment setup. Participants will be randomized to either the intervention or a control group (no active treatment). All participants will be asked to wear a Fitbit Inspire 3 throughout the 8-week study to track physical activity and sleep.

The intervention group will receive access to the MindCo Relief mobile application and a VR headset. The program combining immersive VR mindfulness exercises, cognitive-behavioral education, and self-reflective journaling. Participants may also access up to three optional coaching sessions delivered by trained behavioral health professionals. The control group will complete the same assessments on the same schedule but will not receive any intervention during the study.

Primary and secondary outcomes will be assessed at baseline and 8 weeks post-intervention. The primary outcome is perceived stress (PSS-10). Secondary outcomes include resilience (CD-RISC2), anxiety (GAD-7), depression (PHQ-9), quality of life (GWS), and sleep quality. Hair cortisol will be used to evaluate biological stress response. All survey-based outcomes will be collected online using REDCap.

ELIGIBILITY:
Inclusion Criteria:

* Young adults ages 18-29
* Self-reporting moderate or high perceived stress (PSS-10 score 14 or above)
* able to participate in the trial within 2 weeks after signing informed consent
* have access to a smartphone
* accept to have a hair fragments table for hair cortisol level measurements

Exclusion Criteria:

* Participating in other stress reduction programs
* With photosensitive epilepsy for safety reasons.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2023-10-12 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-05-21 (Actual)

PRIMARY OUTCOMES:
Perceived Stress | From enrollment to the end of treatment at 8 weeks
  Measured by the perceived stress scale 10 Scoring ranges from 0 - 40, and a higher score represents a higher perceived stress. Cutoffs are 0-13 low stress, 14-26 moderate stress, 27-40 high stress

SECONDARY OUTCOMES:
Resilience | From enrollment to the end of treatment at 8 weeks
  Measured by Connor-Davidson Resilience Scale 2 items Scoring ranges from 0 - 8, a higher score represents higher resilience.
Anxiety | From enrollment to the end of treatment at 8 weeks
  General Anxiety Disorder 7 Scoring ranges from 0 - 21, and a higher score represents more severe anxiety. Cutoffs are 0-4 minimal anxiety, 5-9 mild anxiety, 10-14 moderate anxiety, 15-21 severe anxiety.
Depressive symptom | From enrollment to the end of treatment at 8 weeks
  Patient Health Questionnaire - 9
  The scoring ranges from 0 -27, a higher score represents a more severe depressive symptom. Cutoffs are listed below:
  0-4 none-minimal 5-9 mild 10-14 moderate 15-19 moderately severe 20-27 severe
Quality of Life | From enrollment to the end of treatment at 8 weeks
  Measured by general well-being schedule The total score ranges from 0 - 110, with a lower score indicating more severe distress. Cutoffs are 0-60 severe distress, 61-72 moderate distress, 73-110 positive well-being.
Physical activity | From enrollment to the end of treatment at 8 weeks
  Measured by number of steps using Fitbit Inspire 3
Sleep | From enrollment to the end of treatment at 8 weeks
  Sleep data measured by Fitbit Inspire 3
Objective stress | First collection at baseline, second collection at 2 weeks after follow-up assessment was completed
  Measured by hair sample cortisol level

CONTACTS AND LOCATIONS:
Locations (1):
- CUNY SPH, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All data will be available upon reasonable request.